CLINICAL TRIAL: NCT06396871
Title: Deep Phenotyping of Peripheral Blood Cells and Circulating Factors in Metabolic Diseases
Acronym: PERIMED
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: BO-EK-508112022
Record Dates: First submitted 2023-12-22; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: NAFLD; Diabetes Mellitus; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus; Obesity | interventions — Glucose Tolerance Test; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, Serum, Peripheral Blood Mononuclear Cells, Neutrophils, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- High risk - Liver Fibrosis: 1. FIB-4 score ≥ 1.3 AND
  2. Fibroscan measurement ≥ 8kPa
  Interventions: Diagnostic Test: Oral glucose tolerance test; Diagnostic Test: Liver Ultrasound; Diagnostic Test: Fibroscan of the Liver; Diagnostic Test: Magentic Resonance Imaging (MRI) of the liver
- Low risk - Liver Fibrosis: Fibroscan measurements < 8kPa
  Interventions: Diagnostic Test: Oral glucose tolerance test; Diagnostic Test: Liver Ultrasound; Diagnostic Test: Fibroscan of the Liver; Diagnostic Test: Magentic Resonance Imaging (MRI) of the liver
- Steatotic Liver Disease: Diagnosis of steatosis in ultrasound AND CAP > 275 dB/m
  Interventions: Diagnostic Test: Oral glucose tolerance test; Diagnostic Test: Liver Ultrasound; Diagnostic Test: Fibroscan of the Liver; Diagnostic Test: Magentic Resonance Imaging (MRI) of the liver
- No Steatotic Liver Disease: No steatosis in liver ultrasound AND CAP ≤ 275 dB/m
  Interventions: Diagnostic Test: Oral glucose tolerance test; Diagnostic Test: Liver Ultrasound; Diagnostic Test: Fibroscan of the Liver; Diagnostic Test: Magentic Resonance Imaging (MRI) of the liver
- Diabetes: 1. HbA1c ≥ 6.5% OR/AND
  2. Fasting Glucose > 126 mg/dl OR/AND
  3. Glucose at 120 min of OGTT > 200 mg/dl AND/OR history of Diabetes, treated with at least one antidiabetic medication
  Interventions: Diagnostic Test: Oral glucose tolerance test; Diagnostic Test: Liver Ultrasound; Diagnostic Test: Fibroscan of the Liver; Diagnostic Test: Magentic Resonance Imaging (MRI) of the liver
- Prediabetes: 1. HbA1c >5.7 AND <6.5% OR/AND
  2. Fasting Glucose 100-125 mg/dl OR/AND
  3. Glucose at 120 min of OGTT between 140-200 mg/dl
  Interventions: Diagnostic Test: Oral glucose tolerance test; Diagnostic Test: Liver Ultrasound; Diagnostic Test: Fibroscan of the Liver; Diagnostic Test: Magentic Resonance Imaging (MRI) of the liver
- Normal glucose tolerance: 1. HbA1c < 5.7% AND
  2. Fasting glucose < 100 mg/dl AND
  3. Glucose at 120 min of OGTT <140 mg/dl and no history of Diabetes
  Interventions: Diagnostic Test: Oral glucose tolerance test; Diagnostic Test: Liver Ultrasound; Diagnostic Test: Fibroscan of the Liver; Diagnostic Test: Magentic Resonance Imaging (MRI) of the liver

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test — 75g of a standardized glucose solution followed by blood draw at 0, 30, 60, 90, 120 min
Diagnostic Test: Liver Ultrasound — A crude assessment of liver status in order to identify the presence of steatosis or not will take place with ultrasound.
Diagnostic Test: Fibroscan of the Liver — FibroScan non-invasively measures the stiffness of the liver by capturing and calculating the speed of a shear wave as it travels through the liver (vibration controlled transient elastography).
Diagnostic Test: Magentic Resonance Imaging (MRI) of the liver — The exact calculation of liver fat with proton density fat fraction will take place with MRI.

SUMMARY:
The goal of this cross-sectional observational study is to to perform a thorough characterization of the quantitative and qualitative differences in peripheral blood cells, and circulating factors (proteins, metabolites, lipids, extracellular vesicles) in different stages of several metabolic diseases (diabetes, obesity, non-alcoholic fatty liver disease) that share common pathophysiological mechanisms and in comparison with adult healthy controls. The main question[s] it aims to answer are:

* Which are the quantitative (number and concentration) and qualtitative (characteristics, functional assays) differences in platelets in patients with metabolic diseases vs subjects without metabolic diseases
* Which are the quantitative (number and concentration) and qualtitative (characteristics, functional assays) differences in leucocytes or circulating molecules in patients with metabolic diseases vs subjects without metabolic diseases

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old

Additional inclusion criteria for case groups:

1. High risk group for significant liver fibrosis

   1. FIB-4 score ≥ 1.3 AND 2. Fibroscan measurement ≥ 8kPa
2. Steatotic Liver Disease group

   1. Diagnosis of steatosis in ultrasound AND CAP > 275 dB/m
3. Prediabetes

   1. HbA1c >5.7 AND <6.5% OR/AND
   2. Fasting Glucose 100-125 mg/dl OR/AND
   3. Glucose at 120 min of OGTT between 140-200 mg/dl
4. Diabetes 1. HbA1c ≥ 6.5% OR/AND 2. Fasting Glucose > 126 mg/dl OR/AND 3. Glucose at 120 min of OGTT > 200 mg/dl

   If a subject does not fulfil the additional criteria for participating in a case group, then he/she will be included in the respective control group which will be:

   A#) Low risk for significant liver fibrosis 1. Fibroscan measurements < 8kPa B#) No steatosis group

   1. No steatosis in liver ultrasound AND CAP ≤ 275 dB/m C#) Normal glucose tolerance test group
   1. HbA1c < 5.7% AND
   2. Fasting glucose < 100 mg/dl AND
   3. Glucose at 120 min of OGTT <140 mg/dl

   Exclusion Criteria:
   1. Diabetes mellitus Typ 1
   2. BMI < 18.5 kg/m2
   3. Transfusion of blood or major bleeding in the last six months
   4. Anaemia with haemoglobin < 9,0 g/dl
   5. Chronic alcohol or drug abuse
   6. Presence of any acute or chronic liver disease apart from non-alcoholic fatty liver disease (i.e. viral, autoimmune or alcoholic hepatitis, haemochromatosis, Morbus Wilson etc.)
   7. Systemic infections (CRP > 1 mg/dl)
   8. Medications that affect blood glucose levels (e.g. antidiabetics [except from the subjects forming the diabetes group], steroids) in the last six months
   9. Medications that affect coagulation (e.g. anticoagulants and antiplatelet agents) in the last six months
   10. Medications that affect immune function (e.g. immunosuppressive drugs) in the last six months
   11. Pregnancy or breastfeeding
   12. Severe psychic disorders
   13. Inability to follow the study protocol
   14. Have any medical condition unsuitable for inclusion in the study, in the opinion of the investigator

   Additional exclusion criteria for MRI:
   1. Pacemaker
   2. Artificial heart valve
   3. Metal prosthesis
   4. Implanted magnetic metal parts
   5. Spirals
   6. Fixed metal dental braces
   7. Acupuncture needle
   8. Insulin pumps
   9. By MRI > 3 Tesla: Tattoos, permanent eyeliner
   10. Claustrophobia or any other condition, such as psychiatric disorder, that in the opinion of the investigator may prevent the participant from following and completing the protocol
   11. Subject dimensions not allowing the performance of MRI

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population will include subjects belonging to one of the 7 investigation groups. The same subject might belong simultaneously to more than one group (i.e. to fibrosis or no fibrosis group, to steatotic liver disease or no steatotic liver disease group and to normal glucose tolerance, prediabetes or diabetes).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative differences in platelets | 1 day
  % of Platelet aggregation
Quantitative differences in platelets | 1 day
  Platelet count in GPt/L

SECONDARY OUTCOMES:
Quantitative differences in leukocytes | 1 day
  Leucocyte count in GPt/L
Quantitative differences in neutrophils | 1 day
  Neutrophil count in GPt/L
Quantitative differences in lymphocytes | 1 day
  Lymphocyte count in GPt/L
Quantitative differences in monocytes | 1 day
  Monocyte count in GPt/L
Qualitative differences in neutrophils in NETosis | 1 day
  % of neutrophils performing NETosis (FACS analysis)
Qualitative differences in neutrophils in phagocytosis | 1 day
  % of neutrophils performing phagocytosis (FACS analysis)
Qualitative differences in monocytes | 1 day
  % of monocytes performing phagocytosis (FACS analysis)
Quantitative differences in Interleukin-6 | 1 day
  Interleukin-6 in pg/ml
Quantitative differences in Interleukin-8 | 1 day
  Interleukin-8 in pg/ml

CONTACTS AND LOCATIONS:
Locations (1):
- University Study Center for Metabolic Diseases, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided
IPD and biospecimens in pseudonymized form might be shared with other researchers upon written request.